CLINICAL TRIAL: NCT01908647
Title: Using Real-Time Functional Brain Imaging to Enhance Recovery From TBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Van Boven, Robert W., M.D. (Other)
Collaborators: The Geneva Foundation (Other); Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: W81XWH-11-2-0180
Record Dates: First submitted 2013-07-22; First posted 2013-07-26 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Traumatic Brain Injury; Post Traumatic Stress Disorder
Keywords: mTBI; PTSD
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Exp RT fMRI/Exp Cognitive Training (Experimental): Both experimental conditions.
  Interventions: Behavioral: RT fMRI; Behavioral: Cognitive Training
- Exp RT fMRI/Ctrl Cognitive training (Experimental): Experimental real-time fMRI and control cognitive training.
  Interventions: Behavioral: RT fMRI; Behavioral: Control Cognitive Training
- Ctrl RT fMRI/Exp Cognitive Training (Experimental): Control RT fMRI (real-time functional MRI) and experimental cognitive training.
  Interventions: Behavioral: Cognitive Training; Behavioral: Control RT fMRI
- Ctr RT fMRI/Ctr Cognitive Training (Sham Comparator): Control real-time fMRI and control cognitive training.
  Interventions: Behavioral: Control RT fMRI; Behavioral: Control Cognitive Training

INTERVENTIONS:
Behavioral: RT fMRI — Real-time fMRI with neurofeedback.
  Other Names: Real-time fMRI
  Arms: Exp RT fMRI/Ctrl Cognitive training; Exp RT fMRI/Exp Cognitive Training
Behavioral: Cognitive Training — Computer based attention training.
  Arms: Ctrl RT fMRI/Exp Cognitive Training; Exp RT fMRI/Exp Cognitive Training
Behavioral: Control RT fMRI — Control condition for real-time fMRI.
  Arms: Ctr RT fMRI/Ctr Cognitive Training; Ctrl RT fMRI/Exp Cognitive Training
Behavioral: Control Cognitive Training — Computer-based games used as a control for the computer based cognitive training intervention.
  Arms: Ctr RT fMRI/Ctr Cognitive Training; Exp RT fMRI/Ctrl Cognitive training

SUMMARY:
In this randomized, controlled clinical trial, we will evaluate the effects of (1) a brain-training program that uses real-time neurofeedback in functional magnetic resonance imaging (fMRI) to allow people to learn how to gain voluntary control over activity in targeted brain regions and/or (2) 8 weeks of computer-based cognitive training using a software program (Cognitive Remediation for Brain Injury (CRBI)) versus control training tasks on cognitive learning and symptoms. In addition, the investigators will measure brain function (active and resting functional magnetic resonance imaging) and structure (high resolution magnetic resonance imaging) before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Mild TBI: PTA/confusion≤1 hour immediately after injury; or LOC <30 min [69] confirmed by the Ohio confirmed by the Ohio State University TBI Identification Method-Short Form (OSU TBI-ID-SF).
* Age 18-45 years
* Right handed [70].
* Minimum of 4 months and within 36 months post-injury
* Can participate in fMRI and outcome assessment
* Adequate visual, auditory, sensory-motor function for training program.
* Fluent in English
* Persistent cognitive dysfunction confirmed by an objective measure

Exclusion Criteria:

* History of hypoxic event
* Pre-existing significant neurological (e.g. MS) or psychiatric (e.g. schizophrenia, bi-polar) disorders.
* Current illicit drug use or ETOH abuse
* Contraindications to MRI (metal, pregnant, pacemaker, claustrophobia, etc.).
* Unwilling or unable (e.g. language barrier) to participate
* Hospitalization during study
* Current Med Board for discharge, Litigation/ + malingering test [71]
* Use of medications to enhance cognitive function (e.g. Ritalin)
* Initial Glascow Coma Score <13 or penetrating head injury
* Subjects must not show suicidal ideation as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS; 111). Subjects with a score of 4 or 5 (as recommended by the FDA for treatment trials) will be excluded and referred for appropriate treatment.
* Subjects should not be enrolled in a concurrent TBI clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological assessments | 8 weeks
  A composite score based on four primary domains (learning, memory, working memory and executive function).

SECONDARY OUTCOMES:
Participant-reported outcomes | 8 weeks
  A measure of the impact of program use on the participants' own view of their impairment and function
Working/School Status | 8 weeks
  A measure of participants' employment status, schooling status, and the number of hours worked/volunteered/in school per week
Exercise Based Assessments | 4 and 8 weeks
  Three sets of assessments that are closely modeled on study-related exercises in the auditory, visual, and cognitive control modules, and include auditory speed of processing, visual speed of processing, and cognitive control speed of processing.
Functional Assessments | 8 weeks
  Two types of functional measures: a sensitive directly observed performance measure designed originally for normal cognitive aging (timed instrumental activities of daily living, TIADL), and a well-accepted clinical impression measure (the Mayo-Portland Adaptability Inventory, MPAI-4).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Van Boven, M.D., Principal Investigator — The Geneva Foundation
Locations (1):
- Carl R Darnall Army Medical Center (CRDAMC), Fort Hood, Texas, United States